CLINICAL TRIAL: NCT02790437
Title: A Phase II Study to Evaluate the Efficacy of IdeS (IgG Endopeptidase) to Desensitize Transplant Patients With a Positive Crossmatch Test
Brief Title: A Phase II Study to Evaluate the Efficacy of IdeS to Desensitize Transplant Patients With a Positive Crossmatch Test
Acronym: Highdes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hansa Biopharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-HMedIdeS-06
Record Dates: First submitted 2016-05-30; First posted 2016-06-03 (Estimated); Results first posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-04

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment IdeS (Experimental): IdeS intravenous infusion
  Interventions: Drug: IdeS; Procedure: Kidney transplantation

INTERVENTIONS:
Drug: IdeS — One dose of 0.25 mg/kg BW IdeS on study day 0. If negative crossmatch is not achieved, a second dose can be given within 2 days of the first infusion.
  Other Names: IgG endopeptidase
Procedure: Kidney transplantation — Performed following IdeS treatment

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the study drug IdeS in patients who are on the waiting list for kidney transplant and have previously undergone desensitization unsuccessfully or in whom effective desensitization will be highly unlikely. At study entry, the patients will have an available deceased or live donor with a positive crossmatch test. The study will assess IdeS efficacy and safety in removing Donor Specific Antibodies (DSAs) and thereby convert a positive crossmatch test to negative.

DETAILED DESCRIPTION:
The study will assess the IdeS efficacy in creating a negative crossmatch test (XM) in patients who exhibit donor specific antibodies (DSA) and have a positive crossmatch test to their available live or deceased donors. The first 3 patients in this study will receive a kidney from a deceased donor. The study will primarily examine the efficacy of IdeS in creating a negative XM. The first 3 patients will receive one dose of 0.25 mg/kg BW IdeS on study day 0. If it is considered safe and negative crossmatch test is not achieved after the first dose, an additional IdeS infusion can be given within 2 days of the first infusion. The dose schedule may be increased to 0.5 mg/kg BW given once or twice after the first 3 patients have been tested. The decision to escalate the dose will be done after evaluation of safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients on the kidney transplant waitlist who have previously undergone desensitization unsuccessfully or in whom effective desensitization will be highly unlikely. The breadth and strength of sensitization will predict an extremely low likelihood of successful desensitization or kidney paired donation.
* Patients with a live or deceased donor with a positive crossmatch test.

Exclusion Criteria:

* Previous treatment with IdeS
* Previous high dose IVIg treatment (2 g/kg BW) within 28 days prior to IdeS treatment
* Lactating or pregnant females
* Women of child-bearing age who are not willing or able to practice FDA-approved forms of contraception
* HIV-positive patients
* Patients with clinical signs of HBV or HCV infection
* Patients with active tuberculosis
* A significantly abnormal general serum screening lab result according to the investigator's judgement. Hgb cannot be < 6.0 g/dL
* Severe other conditions requiring treatment and close monitoring, e.g. cardiac failure > NYHA (New York Heart Association) grade 3, unstable coronary disease or oxygen dependent COPD
* Individuals deemed unable to comply with the protocol
* Patients with clinical signs of CMV or EBV infection
* Patients with a history of major thrombotic events, patients with active peripheral vascular disease or patients with proven hypercoagulable conditions
* Patients should not have received investigational drugs within 4 half-lives (or similar)
* Known allergy/sensitivity to IdeS infusions
* Patients who have a live donor and test positive for ImmunoCap anti-IdeS IgE

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-06; Primary Completion 2017-12-12 (Actual); Study Completion 2018-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lena Winstedt, PhD, Study Director — Hansa Biopharma AB
Locations (5):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - New York University School of Medicine, New York, New York
- Necker Hospital, Paris, France
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lorant T, Lonze BE, Montgomery RA, Desai NM, Legendre C, Lundgren T, von Zur-Muhlen B, Vo AA, Sjoholm K, Runstrom A, Tollemar J, Jordan SC. Five Years Follow-up of Imlifidase Desensitized Kidney Transplant Recipients. Transpl Int. 2025 Nov 27;38:15425. doi: 10.3389/ti.2025.15425. eCollection 2025. PMID 41394519
- [Derived] Jaffe IS, Runstrom A, Tatapudi VS, Weldon EP, Deterville CL, Dieter RA, Montgomery RA, Lonze BE, Mangiola M. Clinical Outcomes and Donor-specific Antibody Rebound 5 y After Kidney Transplant Enabled by Imlifidase Desensitization. Transplant Direct. 2025 Jan 9;11(2):e1752. doi: 10.1097/TXD.0000000000001752. eCollection 2025 Feb. PMID 39802198
- [Derived] Kjellman C, Maldonado AQ, Sjoholm K, Lonze BE, Montgomery RA, Runstrom A, Lorant T, Desai NM, Legendre C, Lundgren T, von Zur Muhlen B, Vo AA, Olsson H, Jordan SC. Outcomes at 3 years posttransplant in imlifidase-desensitized kidney transplant patients. Am J Transplant. 2021 Dec;21(12):3907-3918. doi: 10.1111/ajt.16754. Epub 2021 Jul 19. PMID 34236770
- [Derived] Jordan SC, Legendre C, Desai NM, Lorant T, Bengtsson M, Lonze BE, Vo AA, Runstrom A, Laxmyr L, Sjoholm K, Schiott A, Sonesson E, Wood K, Winstedt L, Kjellman C, Montgomery RA. Imlifidase Desensitization in Crossmatch-positive, Highly Sensitized Kidney Transplant Recipients: Results of an International Phase 2 Trial (Highdes). Transplantation. 2021 Aug 1;105(8):1808-1817. doi: 10.1097/TP.0000000000003496. PMID 33093408

RESULTS

PARTICIPANT FLOW:
Groups:
- One Dose of IdeS (0.25 mg/kg BW): One (1) IdeS intravenous infusion
  IdeS: One dose of 0.25 mg/kg BW IdeS on study day 0.
  Kidney transplantation: Performed following IdeS treatment
- Two Doses of IdeS (2 x 0.25 mg/kg BW): Two (2) IdeS intravenous infusions
  IdeS: First dose of 0.25 mg/kg BW IdeS on study day 0. Second dose of 0.25 mg/kg BW within 2 days of the first infusion.
  Kidney transplantation: Performed following IdeS treatment
Period: Overall Study
Arm/Group | One Dose of IdeS (0.25 mg/kg BW) | Two Doses of IdeS (2 x 0.25 mg/kg BW)
Started | 16 | 3
Completed | 13 | 3
Not Completed | 3 | 0
Not completed — Patient graft failure - nephrectomy | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- One Dose of IdeS (0.25 mg/kg BW): IdeS: One dose of 0.25 mg/kg BW IdeS on study day 0.
  Kidney transplantation: Performed following IdeS treatment
- Total: Total of all reporting groups
Arm/Group | One Dose of IdeS (0.25 mg/kg BW) | Two Doses of IdeS (2 x 0.25 mg/kg BW) | Total
Number analyzed (Participants) | 16 | 3 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 3 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 40 [20 to 64] | 45 [39 to 45] | 40 [20 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 11 | 2 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 1
  Black or african american | 2 | 2 | 4
  Hispanic | 1 | 0 | 1
  Indian | 1 | 0 | 1
  White | 11 | 1 | 12
Region of Enrollment [Number; unit: participants]
  Sweden | 1 | 1 | 2
  United States | 12 | 2 | 14
  France | 3 | 0 | 3
Weight [Median (Full Range); unit: kg] | 74.05 [45.1 to 107.4] | 68.0 [62.6 to 70.3] | 71.6 [45.1 to 107.4]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Crossmatch Conversion (Positive to Negative)
Description: IdeS ability to create a negative crossmatch (XM) test in patients who before treatment exhibit Donor Specific Antibodies (DSAs) and have a positive XM test to their available live or deceased donor kidney.
  XM was assessed using both FACS and CDC XM tests. FACS XM is a multi-staining procedure where the recipient's serum is used to stain donor cells to identify presence of DSAs in recipient's serum. T- and B-cells are identified using conjugated antibodies against CD3 and CD19. DSAs are identified using a conjugated anti-human antibody. CDC XM evaluates the cytotoxic capacity of the DSAs. The recipient's serum is mixed with donor cells prior to addition of complement. Fluorescent dyes are added and the live/dead cells (%) is scored using a fluorescent microscope. CDC XM amplified with anti-human globulin is not compatible with imlifidase and should not be used.
  The endpoint was met if at least one XM test was positive pre-dose and the last test within 24 h was negative.
Time Frame: Within 24 hours of IdeS dosing
Population: The full analysis set (FAS) comprises data from all patients in the safety analysis set (SAS) with available post-dose efficacy data. Before analysis it was specified that the analysis set should include all patients combined who had received the planned dose which was defined as 1 administration initially which could be repeated if needed. The single as well as the repeated administration are defined as the only planned dose. Consequently, the results are presented for all patients together.
Measure: Number; unit: Patients
Groups:
- FAS - One or Two Doses of 0.25 mg/kg BW IdeS: IdeS intravenous infusion
  IdeS: One dose of 0.25 mg/kg BW IdeS on study day 0. If negative crossmatch is not achieved, a second dose can be given within 2 days of the first infusion.
  Kidney transplantation: Performed following IdeS treatment
  Full analysis set (FAS) comprises all patients in the safety analysis set (SAS) with available post-dose efficacy data.
Arm/Group | FAS - One or Two Doses of 0.25 mg/kg BW IdeS
Number analyzed (Participants) | 19
Patients
  XM conversion within 24 h | 17
  No XM conversion within 24 h | 2

2. Secondary Outcome: Number of Patients With Donor Specific Antibodies With an MFI Value >3000
Description: Donor specific antibodies (DSA) level at different time points within 180 days after administration of IdeS.
  DSA levels were measured using the single antigen beads (SAB) anti-HLA assay. The levels were determined as mean fluorescence intensity (MFI).
  Positive DSA (i.e. HLA antibodies) were defined as having a MFI value >3000.
Time Frame: Within 180 days after administration of IdeS.
Population: The per protocol (PP) set comprises all patients in the SAS with >1 post dose result. Data excluded for patients with >1 protocol deviation. 1 patient lost the graft D77. Before analysis it was specified that the PP set should include all patients combined who had received the planned dose defined as 1 admin. initially which could be repeated if needed. The single as well as the repeated admin. are defined as the only planned dose. Hence, the results are presented for all patients together.
Measure: Number; unit: Patients with DSA (MFI>3000)
Groups:
- PP - One or Two Doses of 0.25 mg/kg BW IdeS: IdeS intravenous infusion
  IdeS: One dose of 0.25 mg/kg BW IdeS on study day 0. If negative crossmatch is not achieved, a second dose can be given within 2 days of the first infusion.
  Kidney transplantation: Performed following IdeS treatment
  The per protocol (PP) set consists of all patients in the safety analysis set (SAS) who had at least one efficacy endpoint value. Data from patients with one or more major protocol deviations were excluded.
Arm/Group | PP - One or Two Doses of 0.25 mg/kg BW IdeS
Number analyzed (Participants) | 18
Patients with DSA (MFI>3000)
  Pre-dose | 17
  2 h | 7
  6 h | 3
  24 h | 3
  48 h | 3
  96 h | 6
  Day 7 | 9
  Day 14 | 13
  Day 28 | 10
  Day 90: number analyzed (Participants) | 17
  Day 90 | 8
  Day 180: number analyzed (Participants) | 17
  Day 180 | 7

3. Secondary Outcome: Time to Create a Negative CDC Crossmatch Test
Description: Time to create a negative CDC crossmatch (XM) was defined as the first timepoint all CDC XM results were negative.
Time Frame: 2h, 6h, 24h after administration of IdeS.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | FAS - One or Two Doses of 0.25 mg/kg BW IdeS
Number analyzed (Participants) | 9
Participants
  All CDC XM tests negative at 2h | 6
  All CDC XM tests negative already pre-dose | 3

4. Secondary Outcome: Time to Create a Negative FACS Crossmatch Test
Description: Time to create a negative FACS crossmatch (XM) was defined as the first timepoint all FACS XM results were negative.
Time Frame: 2h, 6h, and 24h after administration of IdeS
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | FAS - One or Two Doses of 0.25 mg/kg BW IdeS
Number analyzed (Participants) | 19
Participants
  All FACS XM tests negative at 2h | 8
  All FACS XM tests negative at 6h | 2
  All FACS XM tests negative at 24h | 7
  Remained positive | 2

5. Secondary Outcome: Kidney Function After IdeS Treatment Assessed by eGFR
Description: Estimated glomerular filtration rate (eGFR) was calculated as described by the MDRD equation. eGFR is a measure of kidney function.
  eGFR for a kidney with normal function is 90 mL/min/1.72m2. Kidney disease is characterised by a decreased eGFR value.
Time Frame: Within 180 days after administration of IdeS
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PP - One or Two Doses of 0.25 mg/kg BW IdeS
Number analyzed (Participants) | 18
Participants
  Day 28: eGFR: <30 ml/min/1.72m2 | 5
  Day 28: eGFR: 30-59 ml/min/1.72m2 | 9
  Day 28: eGFR: >60 ml/min/1.72m2 | 4
  Day 90: number analyzed (Participants) | 17
  Day 90: eGFR: <30 ml/min/1.72m2 | 4
  Day 90: eGFR: 30-59 ml/min/1.72m2 | 7
  Day 90: eGFR: >60 ml/min/1.72m2 | 6
  Day 180: number analyzed (Participants) | 17
  Day 180: eGFR: <30 ml/min/1.72m2 | 2
  Day 180: eGFR: 30-59 ml/min/1.72m2 | 11
  Day 180: eGFR: >60 ml/min/1.72m2 | 4

6. Secondary Outcome: Serum IgG Concentration After Administration of IdeS
Description: The patient's immunoglobulin G (IgG) is cleaved by IdeS in two steps. The first cut separates one of the heavy chains from the Fc part, generating so called single-cleaved IgG (scIgG), and the second cut separates the other heavy chain from the Fc part, thus generating one F(ab')2 fragment and one Fc fragment. The IgG concentration measured for this outcome is the sum of intact and scIgG because the assay used cannot discriminate between the two. A decrease in IgG concentration therefore represents complete cleavage of the IgG molecules to Fc and F(ab')2 fragments.
  Please note that intravenous IgG (IVIg) was administered Day 7.
Time Frame: Within 180 days after administration of IdeS.
Population: The Per Protocol (PP) analysis set consists of all patients in the safety set who had at least one efficacy endpoint value. Data from patients with one or more major protocol deviations were excluded.
  At Day 180 data was available for 7 patients receiving one dose and 1 patient receiving two doses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/mL
Groups:
- PP - One Dose of 0.25 mg/kg BW IdeS: One (1) IdeS intravenous infusion
  IdeS: One dose of 0.25 mg/kg BW IdeS on study day 0.
  Kidney transplantation: Performed following IdeS treatment
  Per Protocol (PP) analysis set consists of all patients who had at lease one efficacy endpoint value. Data from patients with one or more major protocol deviations were excluded.
- PP - Two Doses of 0.25 mg/kg BW IdeS: Two (2) IdeS intravenous infusion
  IdeS: Two doses of 0.25 mg/kg BW IdeS on study day 0.
  Kidney transplantation: Performed following IdeS treatment
  Per Protocol (PP) analysis set consists of all patients who had at lease one efficacy endpoint value. Data from patients with one or more major protocol deviations were excluded.
- PP - One or Two Doses of 0.25 mg/kg BW IdeS: IdeS intravenous infusion
  IdeS: One dose of 0.25 mg/kg BW IdeS on study day 0. If negative crossmatch is not achieved, a second dose can be given within 2 days of the first infusion.
  Kidney transplantation: Performed following IdeS treatment
  The Per Protocol (PP) set consists of all patients who had at least one efficacy endpoint value. Data from patients with one or more major protocol deviations were excluded.
Arm/Group | PP - One Dose of 0.25 mg/kg BW IdeS | PP - Two Doses of 0.25 mg/kg BW IdeS | PP - One or Two Doses of 0.25 mg/kg BW IdeS
Number analyzed (Participants) | 15 | 3 | 18
mg/mL
  IgG concentration (pre-dose) | 10.11 (85.92) | 8.35 (55.37) | 9.79 (79.73)
  IgG concentration (2 h) | 1.19 (91.05) | 0.68 (165.87) | 1.08 (100.51)
  IgG concentration (6 h) | 0.55 (83.44) | 0.38 (109.18) | 0.52 (85.49)
  IgG concentration (24 h) | 0.37 (79.14) | 0.15 (42.46) | 0.32 (83.92)
  IgG concentration (48 h) | 0.51 (129.17) | 0.17 (45.57) | 0.43 (132.55)
  IgG concentration (Day 7 before IVIg) | 0.64 (107.44) | 0.2 (96.88) | 0.53 (122.3)
  IgG concentration (Day 7 after IVIg) | 16.52 (49.9) | 18.47 (23.91) | 16.89 (45.05)
  IgG concentration (Day 9) | 15.34 (85.32) | 26.94 (50.82) | 16.85 (83)
  IgG concentration (Day 14) | 13.48 (55.67) | 10.85 (53.42) | 13 (54.34)
  IgG concentration (Day 21) | 10.57 (58.67) | 5.88 (88.3) | 9.58 (66.04)
  IgG concentration (Day 28) | 10.25 (69.85) | 11.53 (66.45) | 10.45 (67.16)
  IgG concentration (Day 64) | 11.91 (71.52) | 7.77 (45.82) | 11.09 (69.02)
  IgG concentration (Day 180): number analyzed (Participants) | 7 | 1 | 8
  IgG concentration (Day 180) | 9.33 (42.58) | 8.99 (0) | 9.28 (39.21)

7. Secondary Outcome: Pharmacokinetics - Cmax (First Dose)
Description: Cmax = Maximum observed plasma concentration of IdeS following dosing (Non-compartmental PK analysis)
Time Frame: Pre-dose to Day 14 after administration of IdeS.
Population: The Per Protocol (PP) analysis set consists of all patients in the safety set who had at least one efficacy endpoint value.
  The concentration vs time profiles for all 18 patients, including the 3 patients who received a second dose, were used to calculate Cmax after first dose. Cmax after the first dose occurred before the second dose was administered.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/mL
Groups:
- PP - One or Two Doses of 0.25 mg/kg BW IdeS: IdeS intravenous infusion
  IdeS: One dose of 0.25 mg/kg BW IdeS on study day 0. If negative crossmatch is not achieved, a second dose can be given within 2 days of the first infusion.
  Kidney transplantation: Performed following IdeS treatment
  Per Protocol (PP) set consists of all patients who had at least one efficacy endpoint value. Data from patients with one or more major protocol deviations were excluded.
Arm/Group | PP - One or Two Doses of 0.25 mg/kg BW IdeS
Number analyzed (Participants) | 18
microgram/mL | 3.95 (25.2)

8. Secondary Outcome: Pharmacokinetics - Cmax (Second Dose)
Description: Cmax = Maximum observed plasma concentration of IdeS following dosing (Non-compartmental PK analysis)
Time Frame: Pre-dose until Day 14 after administration of IdeS
Population: The Per Protocol (PP) analysis set consists of all patients in the safety set who had at least one efficacy endpoint value. Data from patients with one or more major protocol deviations were excluded.
  The 3 patients received their second dose 11-13 hours after the first dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/mL
Arm/Group | PP - Two Doses of 0.25 mg/kg BW IdeS
Number analyzed (Participants) | 3
micrograms/mL | 4.13 (29.4)

9. Secondary Outcome: Pharmacokinetics - Tmax (First Dose)
Description: Tmax = Time point for maximum observed plasma concentration of IdeS following dosing (Non-compartmental PK analysis)
Time Frame: Pre-dose to Day 14 after administration of IdeS
Population: The Per Protocol (PP) analysis set consists of all patients in the safety set who had at least one efficacy endpoint value.
  (The mean result presented refers to the arithmetic mean) The concentration vs time profiles for all 18 patients, including the 3 patients who received a second dose, were used to calculate Tmax for the first dose. Cmax/Tmax for the first dose occurred before the second dose was administered.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PP - One or Two Doses of 0.25 mg/kg BW IdeS
Number analyzed (Participants) | 18
hours | 2.21 (0.31)

10. Secondary Outcome: Pharmacokinetics - Tmax (Second Dose)
Description: Tmax = Time point for maximum observed plasma concentration of IdeS following dosing (Non-compartmental PK analysis)
Time Frame: Pre-dose to Day 14 after administration of IdeS
Population: The Per Protocol (PP) analysis set consists of all patients in the safety set who had at least one efficacy endpoint value. Data from patients with one or more major protocol deviations were excluded.
  The 3 subjects received their second dose 11-13 hours after the first dose. Tmax for the second dose was calculated from the start of the first dose.
  (The mean result presented refers to the arithmetic mean.)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PP - Two Doses of 0.25 mg/kg BW IdeS
Number analyzed (Participants) | 3
hours | 15.98 (5.50)

11. Secondary Outcome: Pharmacokinetics - AUC
Description: AUC = Area under the plasma concentration versus time curve (Non-compartmental PK analysis)
Time Frame: Pre-dose to Day 14 after administration of IdeS.
Population: The Per Protocol (PP) analysis set consists of all patients in the safety set who had at least one efficacy endpoint value. Data from patients with one or more major protocol deviations were excluded.
  Data available for 9 patients only who all received 1 dose of IdeS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/mL
Groups:
- PP - Two Doses of 0.25 mg/kg BW IdeS: Two (2) IdeS intravenous infusions
  IdeS: First dose of 0.25 mg/kg BW IdeS on study day 0. Second dose of 0.25 mg/kg BW within 2 days of the first infusion.
  Kidney transplantation: Performed following IdeS treatment.
  Per Protocol (PP) analysis set consists of all patients who had at lease one efficacy endpoint value. Data from patients with one or more major protocol deviations were excluded.
Arm/Group | PP - One Dose of 0.25 mg/kg BW IdeS | PP - Two Doses of 0.25 mg/kg BW IdeS
Number analyzed (Participants) | 9 | 0
hour*microgram/mL | 156.09 (45.4) |

12. Secondary Outcome: Pharmacokinetics - t1/2
Description: Alpha-t1/2 = Half-life during distribution phase Beta-t1/2 = Half-life during elimination phase Non-compartmental PK analysis
Time Frame: Pre-dose to Day 14 after administration of IdeS.
Population: The Per Protocol (PP) analysis set consists of all patients in the safety set who had at least one efficacy endpoint value. Data from patients with one or more major protocol deviations were excluded.
  Data available for 9 patients only who all received 1 dose of IdeS. (The mean result refers to the harmonic mean.)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PP - One Dose of 0.25 mg/kg BW IdeS | PP - Two Doses of 0.25 mg/kg BW IdeS
Number analyzed (Participants) | 9 | 0
hours
  t1/2 (alpha) | 4.58 (3.85) |
  t1/2 (beta) | 76.30 (42.76) |

13. Secondary Outcome: Pharmacokinetics - CL
Description: CL = Clearance Non compartmental PK analysis
Time Frame: Pre-dose to Day 14
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h/kg
Arm/Group | PP - One Dose of 0.25 mg/kg BW IdeS | PP - Two Doses of 0.25 mg/kg BW IdeS
Number analyzed (Participants) | 9 | 0
mL/h/kg | 1.60 (45.4) |

14. Secondary Outcome: Pharmacokinetics - Vss
Description: Vss = Volume of distribution at steady state Non compartmental PK analysis
Time Frame: Pre-dose to Day 14 after administration of IdeS
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/kg
Arm/Group | PP - One Dose of 0.25 mg/kg BW IdeS | PP - Two Doses of 0.25 mg/kg BW IdeS
Number analyzed (Participants) | 9 | 0
L/kg | 0.14 (26.9) |

15. Secondary Outcome: Pharmacokinetics - Vz
Description: Vz = Volume of distribution during the elimination phase Non compartmental PK analysis
Time Frame: Pre-dose to Day 14 after administration of IdeS.
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/kg
Arm/Group | PP - One Dose of 0.25 mg/kg BW IdeS | PP - Two Doses of 0.25 mg/kg BW IdeS
Number analyzed (Participants) | 9 | 0
L/kg | 0.19 (27.0) |

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for 6 months (i.e., from the timepoint the patient signed the informed consent form (ICF) until end of study, including the follow-up period).
Description: Data on AEs were obtained if spontaneously reported by the patient, if reported in response to an open question from the study personnel or if revealed by observation.
  A treatment emergent adverse event (TEAE) was defined as any AE occurring after the administration of IdeS and within the time of the residual drug effect period (i.e. 30 days after IMP administration).
Groups:
- SAS - One Dose of IdeS (0.25 mg/kg BW): One (1) IdeS intravenous infusion
  IdeS: One dose of 0.25 mg/kg BW IdeS on study day 0.
  Kidney transplantation: Performed following IdeS treatment
  The SAS consists of all patients dosed with any amount of IdeS.
- SAS - Two Doses of IdeS (2 x 0.25 mg/kg BW): Two (2) IdeS intravenous infusions
  IdeS: First dose of 0.25 mg/kg BW IdeS on study day 0. Second dose of 0.25 mg/kg BW within 2 days of the first infusion.
  Kidney transplantation: Performed following IdeS treatment.
  The SAS consists of all patients dosed with any amount of IdeS.
- SAS - All Patients (One or Two Doses of IdeS (0.25 mg/kg BW)): One (1) or two (2) IdeS intravenous infusions.
  IdeS: One dose of 0.25 mg/kg BW IdeS on study day 0. If negative crossmatch is not achieved, a second dose can be given within 2 days of the first infusion.
  Kidney transplantation: Performed following IdeS treatment.
  The SAS consists of all patients dosed with any amount of IdeS.
Arm/Group | SAS - One Dose of IdeS (0.25 mg/kg BW) | SAS - Two Doses of IdeS (2 x 0.25 mg/kg BW) | SAS - All Patients (One or Two Doses of IdeS (0.25 mg/kg BW))
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/3 | 0/19
Serious Adverse Events (participants affected / at risk) | 12/16 | 3/3 | 15/19
Other Adverse Events (participants affected / at risk) | 15/16 | 3/3 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAS - One Dose of IdeS (0.25 mg/kg BW) (N=16) | SAS - Two Doses of IdeS (2 x 0.25 mg/kg BW) (N=3) | SAS - All Patients (One or Two Doses of IdeS (0.25 mg/kg BW)) (N=19)
Axillary vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Transplant failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Weaning failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Blood creatine increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Donor specific antibody present (Investigations) | 1 (1) | 0 (0) | 1 (1)
Transplant rejection (Immune system disorders) | 7 (8) | 2 (2) | 9 (10)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombosis in device (General disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Perinephric abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0) | 2 (3)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAS - One Dose of IdeS (0.25 mg/kg BW) (N=16) | SAS - Two Doses of IdeS (2 x 0.25 mg/kg BW) (N=3) | SAS - All Patients (One or Two Doses of IdeS (0.25 mg/kg BW)) (N=19)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 4 (5) | 0 (0) | 4 (5)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 2 (2)
Hypogammaglobulinaemia (Immune system disorders) | 2 (2) | 2 (2) | 4 (4)
Transplant rejection (Immune system disorders) | 1 (2) | 0 (0) | 1 (2)
Administration site pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Application site pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Application site pruritus (General disorders) | 1 (1) | 0 (0) | 1 (1)
Breakthrough pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (2) | 0 (0) | 1 (2)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 1 (1)
Haemorrhagic cyst (General disorders) | 1 (1) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (5) | 1 (2) | 3 (7)
Pain (General disorders) | 2 (5) | 0 (0) | 2 (5)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 0 (0) | 4 (4)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 3 (3)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (2)
Complications of transplant surgery (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 4 (4)
Delayed graft function (Injury, poisoning and procedural complications) | 7 (7) | 1 (1) | 8 (8)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 2 (3)
Procedural pain (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 3 (4)
Renal lymphocele (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 1 (1) | 3 (3)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Clostridium test positive (Investigations) | 1 (1) | 0 (0) | 1 (1)
Donor specific antibody present (Investigations) | 2 (2) | 1 (1) | 3 (3)
Hepatitis B core antibody positive (Investigations) | 1 (1) | 0 (0) | 1 (1)
Respiratory rate decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Sapovirus test positive (Investigations) | 0 (0) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 3 (4) | 1 (1) | 4 (5)
Urine output decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 2 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Throat lesion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 9 (11) | 2 (4) | 11 (15)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 4 (5) | 0 (0) | 4 (5)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 2 (3) | 6 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Tongue paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (12) | 2 (3) | 9 (15)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 0 (0) | 7 (9)
Dyspepsia (Gastrointestinal disorders) | 5 (7) | 0 (0) | 5 (7)
Flatulence (Gastrointestinal disorders) | 2 (3) | 0 (0) | 2 (3)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7) | 1 (1) | 8 (8)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Perianal erythema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (9) | 0 (0) | 7 (9)
Acute kidney injury (Renal and urinary disorders) | 4 (5) | 0 (0) | 4 (5)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal cyst haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (8) | 0 (0) | 6 (8)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 2 (3)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 4 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperparathyroidism secondary (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 3 (3)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 4 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (6) | 2 (4) | 7 (10)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 (5) | 3 (3) | 7 (8)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 4 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (8) | 3 (5) | 9 (13)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 4 (4)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Magnesium deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 7 (7)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (2) | 1 (2)
Perinephric abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pyuria (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (4) | 0 (0) | 2 (4)
Viraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the study, one or more manuscripts for joint publication may be prepared in collaboration between the investigator(s) offered authorship and Hansa Medical AB.

Any confidential information relating to the IMP or the study, including any data and results from the study will be the exclusive property of Hansa Medical AB. The investigator and any other persons involved in the trial will protect the confidentiality of the proprietary information belonging to Hansa Medical AB.

DOCUMENTS (2):
  • Study Protocol (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT02790437/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT02790437/SAP_001.pdf